CLINICAL TRIAL: NCT05986968
Title: Safety of Ticagrelor Monotherapy After Primary Percutaneous Coronary Intervention for ST-elevation Myocardial Infarction and the Effect on Intramyocardial Haemorrhage
Acronym: STOP-IMH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL82646.091.22
Record Dates: First submitted 2023-07-10; First posted 2023-08-14 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Ticagrelor monotherapy instead of dual antiplatelet therapy (aspirin plus ticagrelor)
  Interventions: Drug: Ticagrelor
- Control arm (Active Comparator): Dual antiplatelet therapy (aspirin plus ticagrelor) for 12 months.
  Interventions: Drug: Ticagrelor; Drug: Aspirin

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor monotherapy for 12 months
Drug: Aspirin — Dual antiplatelet therapy (aspirin plus ticagrelor) for 12 months
  Arms: Control arm

SUMMARY:
The main goal of this clinical trial is to assess whether direct omission of aspirin after Percutaneous Coronary Intervention (PCI) with the continuation of ticagrelor monotherapy for 12 months versus 12 months ticagrelor plus aspirin is equally safe regarding the incidence of ischemic events in patients with ST elevation myocardial infarction (STEMI). Furthermore, the two treatment strategies will be compared regarding the incidence and extent of intramyocardial haemorrhage (IMH) and infarct size in the first week after PCI as determined with Cardiac Magnetic Resonance (CMR). The secondary efficacy endpoint consists of clinical bleeding events and all-cause mortality. The main analyses will comprise of clinical outcomes in the first three months after primary PCI and of CMR results. In addition, we will report on clinical outcomes at thirteen months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and electrocardiographical diagnosis of STEMI
* Successful PCI (according to the treating physician) of the infarct-related vessel with a modern drug-eluting stent (DES)

Exclusion Criteria:

* Known allergy or contraindication for aspirin, ticagrelor or prasugrel.
* Previous PCI or MI less than 12 months ago
* Previous cardiac surgery
* Participation in another clinical cardiology study or study concerning platelet aggregation/ thrombosis. (unless the antithrombotic therapy prescribed in this other study will end due to clinical reasons (e.g. the STEMI))
* Pregnancy and breast feeding
* Concurrent use of oral anticoagulants (OAC)
* The periprocedural use of GPIIb/IIIa inhibitors
* Planned surgical intervention within 12 months of PCI
* Creatinine clearance <30mL/min or dialysis
* PCI of stent thrombosis
* Suboptimal stent result as judged by the interventional cardiologist.
* Life expectancy shorter than 13 months.
* Contra-indications for MRI or unable to undergo MRI (only applicable for the CMR subgroup population).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite of major adverse cardiac and cerebral events (MACCE) | 1, 3 and 13 months after primary PCI
  Consisting of: myocardial infarction, stent thrombosis, ischemic stroke, cardiovascular mortality / all-cause mortality
Intramyocardial haemorrhage (IMH) | day 5-8 post primary PCI
  Size of IMH and infarct determined by Cardiac Magnetic Resonance imaging at day 5-8 post primary PCI.

SECONDARY OUTCOMES:
Bleeding complications | 1, 3 and 13 months after primary PCI
  Defined as Bleeding Academic Research Consortium (BARC) 2 or greater
All-cause mortality | 1, 3 and 13 months after primary PCI
Platelet reactivity | 5-8 days
  Differences in platelet reactivity between ticagrelor monotherapy and ticagrelor + aspirin will be measured as Aspirin Reaction Units (ARU) using the VerifyNow test.

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Noordwest Ziekenhuisgroep Alkmaar, Alkmaar
  - Amsterdam UMC, Amsterdam
  - Rijnstate, Arnhem
  - Medisch Spectrum Twente, Enschede
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No